CLINICAL TRIAL: NCT05461404
Title: Emollient Therapy for Improved Survival and Growth of Very Low Birth Weight Infants in Zimbabwe
Brief Title: Emollient Therapy for Premature Infants in Zimbabwe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Collaborators: University of Zimbabwe (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Gary Darmstadt, Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 66546
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Very Low Birth Weight Infant
Keywords: emollient therapy; sunflower seed oil (SSO); skin barrier; Zimbabwe; neonatal mortality; newborn care; preterm infants; postnatal care; growth

STUDY DESIGN:
Intervention Model Description: Infants will be enrolled after informed consent, stratified by birthweight (700- <1000 g, 1000-1500 g) and randomly allocated 1:1 to the two arms of the trial which will be run in parallel.
Masking Description: Due to the visible nature of the intervention, it is not possible to completely mask allocation; thus, the trial will be open-label. However, study physicians will not have access to patient randomization lists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emollient arm (Experimental): Infants will receive gentle, hygienic whole-body massage by trained nurses (not parents or other family members) with 3g of SSO per kg of body weight - a dose sufficient to saturate the skin - three times daily for the first 14 days and twice daily thereafter during the duration of their stay in the hospital until death, discharge or through day 28 after birth.
  Interventions: Other: Topical Emollient Therapy
- Control arm (No Intervention): Infants in the control group will receive the standard of care for infants in the neonatal care unit, which does not include use of topical emollients or massage (i.e., family members will not be allowed to apply skin care products to their infants), or other particular measures to prevent skin breakdown or to modulate skin barrier function.

INTERVENTIONS:
Other: Topical Emollient Therapy — Application of high-linoleate (>60% linoleic acid) SSO to the epidermis.
  Arms: Emollient arm

SUMMARY:
The purpose of this study is to assess the efficacy of topical emollient treatments in improving neonatal growth and mortality rates.

DETAILED DESCRIPTION:
For infants whose parent/caretaker provides written informed consent, the study nurse coordinator on-site will allocate infants to one of two strata (700- <1000 g or 1000-1500 g). Participants within each stratum will be randomly assigned in a 1:1 ratio to one of two treatment groups: 1) high-linoleate SSO, or 2) standard-of-care treatment without use of topical emollients or massage.

ELIGIBILITY:
Inclusion Criteria:

* infants <72 hours of age
* weigh 700-1500 at birth
* hospitalized at SMCH

Exclusion Criteria:

* infants who are moribund and highly likely not to survive despite any intervention
* significant breaches in their skin barrier
* conditions indicating failure to gain weight
* critically ill (definition below):

  1. Oxygen saturation <88% on oxygen therapy AND ≥2 of the following conditions:
  2. respiratory rate <20 or >100 breaths per minute
  3. apnea requiring bag-mask ventilation
  4. heart rate <100 or >200 beats per minute
* congenital syphilis
* hydrops fetalis
* a life-threatening congenital anomaly or major surgical condition requiring intervention
* generalized skin disease or a structural defect involving >5% body surface area likely to produce a defect in epidermal barrier function

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 520 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare mortality rates for VLBW infants treated with SSO vs. control while hospitalized for up to 28 completed days | Baseline and 28 days
  This will be an intent-to-treat analysis, using the randomization level rather than the received level of intervention.
  To estimate the change in mortality rate, we will use a maximum likelihood approach, operationalized as a logistic model with fixed effects for study arm and strata random effects.

SECONDARY OUTCOMES:
Compare growth rates for VLBW infants treated with SSO vs. control while hospitalized for up to 28 completed days. | Baseline and 28 days
  For the secondary analysis of change in growth rate, the quantity of interest is change in weight over the study period as a proportion of the infant's birthweight (g/kg/day). This secondary analysis will use a maximum likelihood approach to both testing and estimation, operationalized as a linear model with fixed effects for the study arm and strata.

OTHER OUTCOMES:
Estimate a strata specific treatment effect, comparing mortality rates in infants 700- <1000 g or 1000-1500 g treated with SSO vs. control. | Within 6 months of the end of enrollment
  This aim will build upon methods used in the primary analysis. To estimate the change in mortality rate, and allowing the treatment effect to vary by strata, we will use a maximum likelihood approach, operationalized as a logistic model with fixed effects for study arm and strata, as well as an interaction term between study arm and strata.
Use residual inclusion modeling to isolate as much as possible the connection between weight gain and mortality. | Within 6 months of the end of enrollment
  For the exploratory analysis which aims to estimate the change in rate of mortality attributable to the change in weight, we will use an instrumental variable design. The study's randomization will be the "instrument," the "treatment" will be change in weight, and the "outcome" of interest will be mortality. This exploratory analysis will use a residual inclusion model approach to both testing and estimation, operationalized as a linear model in the first stage of the residual model and a logistic model in the second stage.

CONTACTS AND LOCATIONS:
Overall Officials: Hilda A. Mujuru, MBChB, MMed, MSc, Principal Investigator — University of Zimbabwe
Locations (1):
- Sally Mugabe Central Hospital (SMCH), Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer N, Darmstadt GL, Shahunja KM, Crowther JM, Kendall L, Gibson RA, Ahmed T, Relman DA. Topical emollient therapy with sunflower seed oil alters the skin microbiota of young children with severe acute malnutrition in Bangladesh: A randomised, controlled study. J Glob Health. 2021 Jul 17;11:04047. doi: 10.7189/jogh.11.04047. eCollection 2021. PMID 34386216
- [Background] Darmstadt GL, Mao-Qiang M, Chi E, Saha SK, Ziboh VA, Black RE, Santosham M, Elias PM. Impact of topical oils on the skin barrier: possible implications for neonatal health in developing countries. Acta Paediatr. 2002;91(5):546-54. doi: 10.1080/080352502753711678. PMID 12113324
- [Background] Cleminson J, McGuire W. Topical emollient for preventing infection in preterm infants. Cochrane Database Syst Rev. 2021 May 7;5(5):CD001150. doi: 10.1002/14651858.CD001150.pub4. PMID 33961715
- [Background] Elias PM, Brown BE, Ziboh VA. The permeability barrier in essential fatty acid deficiency: evidence for a direct role for linoleic acid in barrier function. J Invest Dermatol. 1980 Apr;74(4):230-3. doi: 10.1111/1523-1747.ep12541775. PMID 7373078
- [Background] Prottey C, Hartop PJ, Black JG, McCormack JI. The repair of impaired epidermal barrier function in rats by the cutaneous application of linoleic acid. Br J Dermatol. 1976 Jan;94(1):13-21. doi: 10.1111/j.1365-2133.1976.tb04336.x. PMID 1252336
- [Background] Darmstadt GL, Badrawi N, Law PA, Ahmed S, Bashir M, Iskander I, Al Said D, El Kholy A, Husein MH, Alam A, Winch PJ, Gipson R, Santosham M. Topically applied sunflower seed oil prevents invasive bacterial infections in preterm infants in Egypt: a randomized, controlled clinical trial. Pediatr Infect Dis J. 2004 Aug;23(8):719-25. doi: 10.1097/01.inf.0000133047.50836.6f. PMID 15295221
- [Background] Kumar V, Kumar A, Mishra S, Kan P, Ashraf S, Singh S, Blanks KJH, Baiocchi M, Limcaoco M, Ghosh AK, Kumar A, Krishna R, Stevenson DK, Tian L, Darmstadt GL; Shivgarh Emollient Research Group. Effects of emollient therapy with sunflower seed oil on neonatal growth and morbidity in Uttar Pradesh, India: a cluster-randomized, open-label, controlled trial. Am J Clin Nutr. 2022 Apr 1;115(4):1092-1104. doi: 10.1093/ajcn/nqab430. PMID 34982820
- [Background] Darmstadt GL, Saha SK, Ahmed AS, Chowdhury MA, Law PA, Ahmed S, Alam MA, Black RE, Santosham M. Effect of topical treatment with skin barrier-enhancing emollients on nosocomial infections in preterm infants in Bangladesh: a randomised controlled trial. Lancet. 2005 Mar 19-25;365(9464):1039-45. doi: 10.1016/S0140-6736(05)71140-5. PMID 15781099
- [Background] Darmstadt GL, Saha SK, Ahmed AS, Ahmed S, Chowdhury MA, Law PA, Rosenberg RE, Black RE, Santosham M. Effect of skin barrier therapy on neonatal mortality rates in preterm infants in Bangladesh: a randomized, controlled, clinical trial. Pediatrics. 2008 Mar;121(3):522-9. doi: 10.1542/peds.2007-0213. PMID 18310201
- [Background] Salam RA, Darmstadt GL, Bhutta ZA. Effect of emollient therapy on clinical outcomes in preterm neonates in Pakistan: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2015 May;100(3):F210-5. doi: 10.1136/archdischild-2014-307157. Epub 2015 Jan 30. PMID 25637007
- [Background] Salam RA, Das JK, Darmstadt GL, Bhutta ZA. Emollient therapy for preterm newborn infants--evidence from the developing world. BMC Public Health. 2013;13 Suppl 3(Suppl 3):S31. doi: 10.1186/1471-2458-13-S3-S31. Epub 2013 Dec 20. PMID 24564550
- [Background] Kumar A, Mishra S, Singh S, Ashraf S, Kan P, Ghosh AK, Kumar A, Krishna R, Stevenson DK, Tian L, Elias PM, Darmstadt GL, Kumar V; Shivgarh Emollient Research Group. Effect of sunflower seed oil emollient therapy on newborn infant survival in Uttar Pradesh, India: A community-based, cluster randomized, open-label controlled trial. PLoS Med. 2021 Sep 28;18(9):e1003680. doi: 10.1371/journal.pmed.1003680. eCollection 2021 Sep. PMID 34582448
- [Derived] Hui A, Chimhini G, Saungweme M, Kaisi D, Munetsi E, Mujuru HA, Darmstadt GL. Postnatal care and acceptability of emollient therapy in very low birthweight infants in Harare, Zimbabwe: a qualitative analysis. BMC Pediatr. 2024 Mar 16;24(1):187. doi: 10.1186/s12887-024-04661-x. PMID 38493088